CLINICAL TRIAL: NCT00918398
Title: An Open, Single-dose, Phase I, 4-period Partly Crossover Study in Healthy Men or Women to Assess Relative Bioavailability of Oral Administration of AZD1981 Via Tablets Compared With Suspension and Basic Systemic Pharmacokinetic Parameters After Intravenous Administration
Brief Title: AZD1981 Bioavailability Study of Intravenous (IV) and Oral Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist, Medical Science Director, AstraZeneca R&D Lund, Sweden
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D9831C00003; EudraCT No. 2009-010964-40
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Healthy; Postmenopausal; Surgically Sterile Women
MeSH Terms: interventions — AZD1981

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): AZD1981, 100 mg iv infusion
  Interventions: Drug: AZD1981
- 2 (Experimental): AZD1981, 514 mg oral solution
  Interventions: Drug: AZD1981
- 3 (Experimental): AZD1981, 500 mg oral tablet A
  Interventions: Drug: AZD1981
- 4 (Experimental): AZD1981, 500 mg oral tablet B
  Interventions: Drug: AZD1981

INTERVENTIONS:
Drug: AZD1981 — 100 mg iv infusion, single dose, 4 hours infusion
  Arms: 1
Drug: AZD1981 — 514 mg oral solution, single dose
  Arms: 2
Drug: AZD1981 — 500 mg oral tablet A (optimal dissolution) give as 2x250 mg tablets, single dose
  Arms: 3
Drug: AZD1981 — 500 mg oral tablet B (slower dissolution) give as 2x250 mg tablets, single dose
  Arms: 4

SUMMARY:
The primary objective is to investigate the pharmacokinetics of AZD1981 given in different formulations and to measure renal clearance

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Men or post-menopausal or surgically sterile women, aged 18 to 55 years
* Have a body mass index between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to Visit 1 (pre-entry)

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the result of the study, or the subject´s ability to participate
* Any clinically relevant abnormal findings in phys.examination, clinical chemistry, haematology, urinalysis, vital signs, or ECG at baseline which, in the opinion of the investigator, may put the subject at risk because of his participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2009-06; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
PK samples for AZD1981 from both blood and urine | Intense PK-sampling during the 24 hours following dose and additional samples up to 60 hours after dose.

SECONDARY OUTCOMES:
Safety variables (adverse events and laboratory safety lab) | Adverese events registered during study and vital signs and ECG at visit 1,2 ,6

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pettersson, Study Director — AstraZeneca R&D, Lund, Sweden; Elisabeth Eden, Principal Investigator — Quintiles AB, Uppsala, Sweden
Locations (1):
- Research Site, Uppsala, Sweden